CLINICAL TRIAL: NCT01009021
Title: Analgesic Effectiveness of Potassium Diclofenac for Retinal Photocoagulation in Patients With High-risk Proliferative Diabetic Retinopathy
Brief Title: Oral Diclofenac for Retinal Photocoagulation in Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Rodrigo Jorge, University of Sao Paulo Professor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NSAID-PRP
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Pain
Keywords: pain; retinal photocoagulation; potassium diclofenac
MeSH Terms: conditions — Pain | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo first (scheme 2) (Other): scheme 2 patients (n=15) received a brown-coated tablet of saccharine (placebo) 45 minutes before the first PRP episode [placebo treatment episode (PTE)] at baseline to the right eye and two weeks after received one 50 mg tablet of potassium diclofenac 45 minutes before the second PRP episode [diclofenac treatment episode (DTE)] to the left eye
  Interventions: Drug: potassium diclofenac
- Diclofenac first (scheme 1) (Other): scheme 1 patients (n=15) received one 50 mg tablet of potassium diclofenac 45 minutes before the first PRP episode [diclofenac treatment episode (DTE)] at baseline to the right eye and two weeks after received an identical brown-coated tablet of saccharine (placebo) 45 minutes before the second PRP episode [placebo treatment episode (PTE)] to the left eye
  Interventions: Drug: potassium diclofenac

INTERVENTIONS:
Drug: potassium diclofenac — potassium diclofenac 50 mg, one tablet 45 minutes before laser treatment
  Other Names: Cataflan

SUMMARY:
The purpose of this study was to evaluate the analgesic effect of oral potassium diclofenac in patients with proliferative diabetic retinopathy submitted to retinal photocoagulation.

Two groups of patients were followed and the effect of the treatment (diclofenac plus laser) was compared to placebo (placebo plus laser). Pain associated with treatment was recorded using a Visual Analog Scale 15 minutes after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 1)high-risk proliferative diabetic retinopathy in both eyes

Exclusion Criteria:

* 1)history of prior laser treatment or vitrectomy; 2) allergy to non-steroidal anti-inflammatory drugs; 3) any condition affecting comprehension of VAS pain score test; 4) Contra-indications for diclofenac use such as pregnancy, bleeding disorders, asthma, or renal failure; 5) use of any analgesic drug for the last 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain recorded using a Visual Analog Scale | 15 minutes after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Ribeirão Preto School of Medicine Clinics Hospital - USP, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Lucena CR, Ramos Filho JA, Messias AM, Silva JA, Almeida FP, Scott IU, Ribeiro JA, Jorge R. Panretinal photocoagulation versus intravitreal injection retreatment pain in high-risk proliferative diabetic retinopathy. Arq Bras Oftalmol. 2013 Jan-Feb;76(1):18-20. doi: 10.1590/s0004-27492013000100006. PMID 23812521